CLINICAL TRIAL: NCT04487639
Title: Presence of SARS-CoV-2 in Semen: Impact on Fertility Preservation in Male Oncological Patients During the COVID-19 Pandemic ?
Brief Title: Presence of SARS-CoV-2 (COVID-19) in Semen: Impact on Fertility Preservation in Male Oncological Patients ?
Acronym: FERTICOVID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Agence de La Biomédecine (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RNI 2020 BRUGNON; 2020-A01409-30 (Other: ANSM)
Record Dates: First submitted 2020-07-21; First posted 2020-07-27 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Sperm Preservation in Oncological Patients; Fertility; Cryopreservation
Keywords: Fertility preservation; Sperm; Cancer; COVID-19; SARS-CoV-2
MeSH Terms: conditions — Neoplasms; COVID-19 | interventions — Sperm Count

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cohort : patients needing oncofertility preservation (Experimental)
  Interventions: Diagnostic Test: SARS-CoV-2 research in nasopharyngeal swab, sperm and serologics

INTERVENTIONS:
Diagnostic Test: SARS-CoV-2 research in nasopharyngeal swab, sperm and serologics — a nasopharyngeal swab for SARS-CoV-2 research by RT- qPCR will be performed on the day of semen collection. On the same day, serological tests will be carried out, and 30 to 50 days after, according to HAS specifications with methods validated by the National Reference Center

SUMMARY:
During the COVID-19 pandemic, the French Agency of Biomedicine has recommended maintaining fertility preservation for patients requiring immediate oncological treatments exhibiting gonadotoxic effects. However, no study has examined the presence of SARS-CoV-2 in sperm from cancer patients. This study aims therefore to detect the presence of SARS-CoV-2, specifically in the seminal fluid and the spermatozoa fractions of cancer patient semen. The investigators will determine if the virus presence in sperm is associated with its presence in the nasal swabs, COVID symptoms, specific serological profiles and particular oncological pathologies/treatments.

DETAILED DESCRIPTION:
To perform this, all patient undergoing oncological fertility preservation will be evaluated for COVID-19 symptomatology (fever, cough, headache, myalgia, diarrhea, anosmia, pharyngodynia). In addition, a nasopharyngeal swab for SARS-CoV-2 research by RT- qPCR will be performed on the day of semen collection. On the same day, serological tests will be carried out, and 30 to 50 days after, according to HAS specifications with methods validated by the National Reference Center. Seminal fluid and spermatozoa will be separated by density gradient centrifugation for a posteriori molecular analysis of SARS-CoV-2 presence.

Will thus be measured, within the same ejaculate, the concordance between the presence of SARS-CoV-2 in the seminal fluid and in the sperm cells fraction.

The investigators will also determine if the virus presence in the sperm is related with :

* (i) the presence of SARS-CoV-2 in the nasal swab;
* (ii) patient symptomatology;
* (iii) a specific serological profile;
* (iv) a particular oncological pathology and / or treatment. The investigators may also find out if the presence of the SARS-CoV-2 in semen affects sperm quality.

This study will be the first one examining the presence of SARS-CoV-2 in semen from cancer patients. This will guarantee the safety of fertility preservation procedures during the COVID-19 pandemic.

ELIGIBILITY:
Inclusion Criteria:

* Man above 18 years of age, of reproductive age, needing oncofertility preservation through spermatozoa cryopreservation prior to a putative gonadotoxic treatment during the COVID-19 pandemic.
* Symptomatic and asymptomatic COVID-19 patients. A patient is considered as symptomatic if he presents one or several of the following clinical signs: fever, cough, cephalalgia, myalgia, diarrhea, anosmia, pharyngodynia.
* A sufficient number of remaining spermatozoa straws to perform at least six ART attempts

Exclusion Criteria:

* Azoospermia
* Severe Oligo-Astheno-Teratozoospermia (OAT) or Cryptozoospermia
* Semen collection failure
* Non-emergency fertility preservation or treatment with low gonadotoxic risk

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 129 (Actual)
Dates: Start 2020-07-10 (Actual); Primary Completion 2021-07-02 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Detection of SARS-CoV-2 in sperm during fertility preservation procedures by RT-qPCR | Semen collection day (Day0)
  Seminal fluid and spermatozoa will be separated by density gradient centrifugation, and SARS-CoV-2 will be detected by RT-qPCR in the both fractions.

SECONDARY OUTCOMES:
To correlate the presence of SARS-CoV-2 in the seminal fluid and the spermatozoa fractions of the same ejaculate | Semen collection day (Day0)
  We will compare SARS-CoV-2 RT-PCR results of seminal fluid and the spermatozoa fractions of the same ejaculate
To determine if the presence of this virus in sperm is associated with its presence in nasal swabs | Semen collection day (Day0)
  we will correlate the SARS-CoV-2 detection (using RT- qPCR) in nasopharyngeal swab, seminal fluid and spermatozoa fractions
To determine if the presence of this virus in sperm is associated with COVID symptoms | Semen collection day (Day0)
  Any patient undergoing oncological fertility preservation will be evaluated for COVID-19 symptomatology (fever, cough, headache, myalgia, diarrhea, anosmia, pharyngodynia). We will correlate the SARS-CoV-2 detection in seminal fluid and spermatozoa fractions with COVID symptoms
To determine if the presence of this virus in sperm is associated with specific serological profiles | Semen collection day (Day0) and 30 to 50 days after (Day 30 to 50)
  Serological tests (Sars-CoV2) will be carried out. We will correlate the SARS-CoV-2 detection in seminal fluid and spermatozoa fractions with specific COVID serological profiles
To determine if the presence of this virus in sperm is associated with particular oncological pathologies/treatments | Semen collection day (Day0)
  We will correlate the SARS-CoV-2 detection in seminal fluid and spermatozoa fractions with patient's oncological pathologies and treatments
To determine if the presence of this virus in sperm could impair its quality | Semen collection day (Day0)
  Before semen density gradient centrifugation and cryopreservation, standards sperm analysis will be performed according to the WHO guideline (2020). We will correlate the SARS-CoV-2 detection in seminal fluid and spermatozoa fractions with standards sperm parameters

CONTACTS AND LOCATIONS:
Overall Officials: Florence BRUGNON, MD, PhD, Principal Investigator — CHU de Clermont-Ferrand
Locations (16):
- France (16):
  - AP-Hôpitaux de Paris - Hôpital Jean Verdier - Service de Biologie de la reproduction, Bondy
  - AP-Hôpitaux de Paris - Hôpital Antoine Béclére - Service de Biologie de la reproduction et AMP DPI CECOS, Clamart
  - CHU de Clermont-Ferrand - Laboratoire de Virologie, Clermont-Ferrand
  - CHU de Clermont-Ferrand, Clermont-Ferrand
  - CHU de Dijon - Laboratoire de Biologie de la Reproduction-CECOS, Dijon
  - CHU de Grenoble - Laboratoire d'Aide à la Procréation CECOS, Grenoble
  - Hospices Civils de Lyon - Service AMP-CECOS, Lyon
  - Hôpital de la Conception - AP-Hôpitaux de Marseille - Service AMP-CECOS, Marseille
  - CHU de Nancy - Laboratoire de biologie de la reproduction - CECOS, Nancy
  - AP-Hôpitaux de Paris - Hôpital Tenon - Service de Biologie de la reproduction - CECOS, Paris
  - AP-Hôpitaux de Paris - Hôpital Cochin - Service d'Histologie-Embryologie-Biologie de la reproduction, Paris
  - Centre Hospitalier intercommunal (CHI) de Poissy Saint Germain en Laye, Poissy
  - CHU de Reims - Service de Biologie de la Reproduction - CECOS Champagne-Ardenne de Reims, Reims
  - CHU de Rouen Normandie - Service Biologie de la Reproduction-CECOS, Rouen
  - CHU de Strasbourg - Service de Biologie de la reproduction, Strasbourg
  - CHU de Toulouse - CECOS Midi-Pyrénées, Toulouse

IPD SHARING:
Plan to Share IPD: No